CLINICAL TRIAL: NCT06666634
Title: Validation of ICG-99mTc-nanoscan as Hybrid Tracer for Sentinel Node Biopsy
Acronym: NANOSCAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N21NAN
Record Dates: First submitted 2023-03-01; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Penile Cancer; Melanoma; Oral Cancer
Keywords: Fluorescence; Radioactivity; Indocyanine green; Clinical node negative patients; Surgical staging
MeSH Terms: conditions — Penile Neoplasms; Melanoma; Mouth Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dynamic sentinel node biopsy with 99mTc-nanoscan and ICG-99mTc-nanoscan (Other): The patient first receives a one-time injection with 99mTc-nanoscan, then a one-time injection with ICG-99mTc-nanoscan, both dosage are according to routine care.
  Interventions: Drug: Sentinel node biopsy with either ICG-99mTc-nanoscan or 99mTc-nanoscan

INTERVENTIONS:
Drug: Sentinel node biopsy with either ICG-99mTc-nanoscan or 99mTc-nanoscan — Sentinel node biopsy with either ICG-99mTc-nanoscan or 99mTc-nanoscan

SUMMARY:
99mTc-nanocolloid, the world wide used hybrid tracer for dynamic sentinel node biopsy, has recently been replaced with 99mTc-nanoscan. The hybrid form (ICG-99mTc-nanoscan) has not yet been validated, to show the similarity between the lymphatic drainage pattern between ICG-99mTc-nanoscan and 99mTc-nanoscan.

DETAILED DESCRIPTION:
The investigators want to set up this study in analogy with the comparison study which was conducted before the introduction of ICG-99mTc-Nanocolloid (99mTc-Nanocoll vs. ICG-99mTc-Nanocoll (NL26699.031.09 -N09DRF). In particular, the investigators want to validate that the hybrid ICG-99m Tc-Nanoscan shows the same preoperative gland involvement on preoperative lymphoscintigraphy and that the intraoperative signal intensities remain the same. All this to maintain the level of current care.

ELIGIBILITY:
Inclusion Criteria:

* Patient who will undergo a sentinel node procedure in routine care.
* Patients > 18 years;
* Patients presenting with:
* a primary cutaneous melanoma of head/neck or upper part of the trunk or extremities;
* OR patients presenting with a primary oral cavity malignancy T1-2N0
* OR patients with primary penile cancer
* Patients with clinical N0 stage;
* Patients scheduled for a sentinel node biopsy prior to (re-)excision of the primary lesion;
* Patients in which ICG-99mTc-nanoscan would be used in routine care or a research setting

Exclusion Criteria:

* Patients with known allergy to patent blue dye or nanocolloid;
* Patients who are pregnant or breast-feeding mothers;
* History of hypersensitivity reactions to products containing human serum albumin;
* History of iodine allergy
* Hyperthyroid or thyroidal adenoma
* Kidney insufficiency
* Incapacity or unwillingness of participant to give written informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Concordance between tracers | Measured at pre-operative imaging
  To demonstrate concordance between the SN visualization of 99mTc-nanoscan and ICG-99mTc-nanoscan on preoperative lymphoscintigraphy and SPECT/CT imaging, expecting an average of 3 sentinel nodes per patient. Discordance is defined as more than 1 sentinel node not detected coherently by the tracers.

SECONDARY OUTCOMES:
Higher echelon nodes | Measured at pre-operative imaging
  Number of higher-echelon nodes visualized on preoperative lymphoscintigraphy and SPECT/CT imaging for both tracers (ICG-99mTc-Nanoscan and 99mTc-Nanoscan);
Concordance between intraoperative fluorescence and radioactive findings | Measured at pre-operative imaging
  Number of the fluorescent nodes at time of excision;
  - Number and radioactive signal intensity of the radioactive nodes at time of excision;
Concordance between intraoperative fluorescence and radioactive findings | Measured at pre-operative imaging
  intensity of the fluorescent nodes at time of excision;

CONTACTS AND LOCATIONS:
Locations (1):
- NKI-AVL, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No